CLINICAL TRIAL: NCT02739399
Title: The Dynamic Effects of Phenylephrine on Preload and Cardiac Output in Patients Under General Anaesthesia
Brief Title: Effects of Phenylephrine on Cardiac Preload
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Dr, Algemeen Ziekenhuis Maria Middelares
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM2015.037
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Arterial Hypotension; Anaesthesia
Keywords: phenylephrine; alpha mimetics; pulse pressure variation; venous return
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient receiving phenylephrine 2ug/kg (Other): phenylephrine 2ug/kg in case of hypotension
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — Intravenous administration
  Other Names: Phenyl

SUMMARY:
In patients under general anesthesia, episodes of hypotension are often treated with phenylephrine. The effect of phenylephrine is conventionally attributed to afterload increase.

The aim of the study is to describe the time course of the effects of phenylephrine on the cardiac preload and cardiac output, and to evaluate whether phenylephrine, as an exclusive alpha-mimetic, could be beneficial for preload optimisation.

DETAILED DESCRIPTION:
In consecutive patients scheduled for laparoscopic sigmoidectomy, all hemodynamic and respiratory variables are recorded electronically for subsequent offline analysis.

All patients are ventilated in volume control mode with a tidal volume of 8 ml/kg ideal body weight.

During steady-state Target Controlled Infusion (TCI) propofol/remifentanil anesthesia, when the Mean Arterial Blood Pressure (MAP) dropped below 80% of the awake state for at least 5 minutes, a phenylephrine bolus of 2 μg/kg is administered. If necessary this is repeated, or a continuous administration of phenylephrine is started at a rate of 10-30 μg/kg/u.

All patient manipulations during the procedure are electronically recorded and time stamped for subsequent off-line data analysis.

The first episode in each patient where phenylephrine is administered and in a period of at least 10 minutes when minimal or absent patient manipulation occurred, the hemodynamic variables are analysed to describe the effects of phenylephrine administration on the dynamic preload parameters and macro-hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* necessity for arterial blood pressure monitoring
* necessity for central venous blood pressure monitoring

Exclusion Criteria:

* unwilling or unable to grant written informed consent
* cardiac arrythmia
* contra-indication for phenylephrine
* contra-indications for atropine
* contra-indication for Total Intravenous Anesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cardiac output | perioperative
  The evolution of the Cardiac Output in a time course <20 minutes after administration

SECONDARY OUTCOMES:
Pulse Pressure Variation | perioperative
  The evolution of Pulse Pressure Variation in a time course <20 minutes
End-Tidal CO2 | perioperative
  The evolution of the EtCO2-value in a time course <20 minutes
Arterial Blood Pressure | perioperative
  The evolution of The Arterial Blood Pressure in a time course <20 minutes
central venous pressure | perioperative
  The evolution of the central venous pressure in a time course <20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD, PhD, Principal Investigator — Department of Anaesthesiology and Intensive care medicine, Maria Middelares hospital, Ghent, Belgium
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No